CLINICAL TRIAL: NCT03614338
Title: A Small Changes Weight Loss Program and Message Dissemination Via Facebook in Chicago's West Side
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Melissa M. Crane, PhD, Assistant Professor, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18070904
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Core Participants Weight Loss Program (Experimental): Small changes weight loss program
  Interventions: Behavioral: Small changes weight loss program

INTERVENTIONS:
Behavioral: Small changes weight loss program — This intervention uses a "small-changes" approach to calorie reduction (operationalized as 6 100-calories changes per day) along with increasing leisure-time physical activity and self-regulation strategies to produce weight loss. The intervention will be delivered via 12 face-to-face group sessions.

SUMMARY:
African-American communities experience a greater burden of obesity-related diseases such as type 2 diabetes mellitus and cardiovascular disease and higher rates of obesity, compared to other race groups. There is a need for interventions that show promise in mitigating these disparities. The primary goal of this project is to pilot test whether an existing "small-changes" intervention for weight loss can be modified and delivered within the West Side ALIVE churches.

ELIGIBILITY:
Inclusion Criteria:

1. BMI 25-45 kg/m2
2. Age 18-75
3. Attend one of the West Side partnership churches at least 2 times per month
4. Able to attend in-person meetings
5. Willing to share their experiences on the West Side ALIVE Facebook page

Exclusion Criteria:

1. Blood pressure > 170/90 (self-report or during the WSA screening)
2. Diabetes treated with insulin
3. History of cancer within the past 5 years
4. Pregnancy or breastfeeding in the last 6 months, planning to become pregnant in the next 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Weight | 3 months
  Change from baseline using objectively measured body weight

SECONDARY OUTCOMES:
Blood pressure | 3 months
  Change from baseline
Physical activity | 3 months
  Change from baseline in total minutes of MVPA assessed by accelerometer
Weight loss strategies | 3 months
  Change from baseline on self-reported use of weight loss strategies
Weight | 6 months
  Change from baseline using objectively measured body weight
HbA1c | 3 months
  Change from baseline using a point of care analyzer

OTHER OUTCOMES:
Program satisfaction | 3 months
  Self-reported program satisfaction post-intervention
Program engagement | 3 months
  Number of sessions attended during intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No